CLINICAL TRIAL: NCT05395169
Title: EFFECT OF DASH DIET AND AEROBIC EXERCISES ON PREMENSTRUAL SYNDROME
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Mabrouk El-Said Anwer, specialist physical therapist at Al Delangat Hospital, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.TREC/012/003692
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Premenstrual Tension
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- medical treatment (Experimental): Control group:Will be consisted of 25 females suffering from PMS will receive medical treatment in form of vit, B6, ca supplements and minerals (vitatron), once daily(1capsule), for 12 weeks.
  Interventions: Other: dietary supplement ,electronic treadmill ,DASH diet.
- the same medication, in addition to DASH diet and aerobic exercise (Experimental): Study group: Will be consisted of 25 females suffering from PMS will Receive the same medication as in group (A) in addition to the DASH diet and aerobic exercise for 30 minutes,3 times/week,for 12 weeks.
  Interventions: Other: dietary supplement ,electronic treadmill ,DASH diet.

INTERVENTIONS:
Other: dietary supplement ,electronic treadmill ,DASH diet. — Control group Will be receive medical treatment for 12 weeks. Study group Will be receive the same medication as in control group in addition to DASH diet and aerobic exercise for 12 weeks.

SUMMARY:
Hypothesis:

There will be no effect of the DASH diet and aerobic exercise on premenstrual syndrome.

Statement of the problem:

Do the DASH diet and aerobic exercise have an effect on premenstrual syndrome?

DETAILED DESCRIPTION:
For some women, symptoms of PMS may be so severe that they miss work or school. Physical activity is a suitable method for the treatment of PMS and is the best method for all women to reduce pressure and balance the brain's chemical secretion. It seems that physical activity by increasing endorphins and reducing adrenal cortisol leads to the improvement of symptoms of PMS.

DASH diet has been suggested to play an important role in the development, and treatment of some psychological disorders. For instance, it has been reported that a diet rich in fish, folate, and B-vitamins can alleviate the manifestations of depression. An established association was also shown between the dietary glycemic index (GI) and psychological diseases, depressive disorder, and mental functioning.

Diets containing of "junk foods" (high energy and low nutritional) have been shown to increase the risk of mental illness, but a healthy diet is associated with less depressive symptoms and can improve mood .

ELIGIBILITY:
Inclusion Criteria:

* Fifty adolescent females were diagnosed with premenstrual syndrome.
* Their age will be ranged from 15-to 25 years (3 years post-puberty).
* Their body mass index (BMI) will range from 18-25.9 kg/m2.
* All are of regular menstrual cycles.
* All of them suffer from moderate and severe PMS.

Exclusion Criteria:

* Any pathologic findings in the pelvic cavity as a polycystic ovarian syndrome, endometriosis, and pelvic inflammatory diseases.
* Having irregular menstruation.
* Any metabolic diseases.
* Any history of gynecological intervention.

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | assessment will be take 12 weeks
  Visual analogue scale (VAS):
  Degrees of menstrual pain will be assessed using a VAS for all participants in both groups (A&B) before and after treatment, which is a method of representing .participants pain on a 10 cm linear scale. A score of zero mean "a very low degree of pain" and 10 mean "a very high degree of pain"
Menstrual Distress Questionnaire (MDQ) | assessment will be take 12 weeks
  Menstrual Distress Questionnaire (MDQ):
  The subjects decreased activity, lower back pain, tension or anxiety, breast tenderness, and headaches will assess for all participants in both group before and after treatment using Menstrual Distress Questionnaire (MDQ) .Each item will be score on a 5-point likert scale ,with 1 being "no pain at all" follow by "mild pain", "moderate pain", "slightly sever pain" ,and "extremely severe pain.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF